CLINICAL TRIAL: NCT02734888
Title: Arterial Inflammation and E-Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Holly R Middlekauff, Professor of Medicine, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-000552
Record Dates: First submitted 2016-04-01; First posted 2016-04-12 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Arterial Inflammation
Keywords: arterial inflammation; electronic cigarettes; PET scan
MeSH Terms: conditions — Arteritis; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy control (Other): Will undergo PET scan as a "negative control"
  Interventions: Other: No drug or device, only a test. The test is called a PET/CT
- Tobacco cigarette smoker (Other): Will undergo PET scan as a "positive control"
  Interventions: Other: No drug or device, only a test. The test is called a PET/CT
- E-cigarette user (Other): Will undergo PET scan
  Interventions: Other: No drug or device, only a test. The test is called a PET/CT

INTERVENTIONS:
Other: No drug or device, only a test. The test is called a PET/CT — A single PET/CT scan will be performed

SUMMARY:
Arterial inflammation will be compared using PET scanning in 3 groups: 1) Non-smokers, 2) Tobacco cigarette smokers, 3) Electronic cigarette users.

DETAILED DESCRIPTION:
Qualified participants will undergo a singe PET/CT to detect arterial inflammation.

ELIGIBILITY:
Inclusion Criteria:

Healthy

* Nonsmokers OR
* Daily e-cigarette user OR
* Daily tobacco cigarette smoker

Exclusion Criteria:

* Cardiac disease
* Respiratory Disease
* Diabetes mellitus

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
target-to-background ratio (TBR) | intraoperative
  TBR will be detected on the scan

CONTACTS AND LOCATIONS:
Overall Officials: Holly R Middlekauff, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCaliforniaLA, Los Angeles, California, United States